CLINICAL TRIAL: NCT07132008
Title: Prospective, Multicenter, Randomized Trial of Neoadjuvant Capecitabine and Oxaliplatin (CAPOX) Plus Tislelizumab Versus CAPOX in Microsatellite Stable High-risk Locally Advanced Colon Cancer
Brief Title: Neoadjuvant CAPOX Plus Tislelizumab vs CAPOX in MSS High-Risk Locally Advanced Colon Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Collaborators: The First Affiliated Hospital of Xiamen University (Other); The First Affiliated Hospital of University of South China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-K0173
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Colonic Neoplasms; Neoadjuvant Therapy; Immune Checkpoint Inhibitors
Keywords: Colon cancer; Neoadjuvant chemotherapy; PD-1 inhibitor
MeSH Terms: conditions — Colonic Neoplasms | interventions — tislelizumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAPOX combined with Tislelizumab (Experimental): Patients in the experimental group underwent two or four cycles of preoperative CAPOX combined with Tislelizumab. Patients assessed as suitable for R0 resection by imaging underwent radical colectomy. Following surgery, all patients in both groups completed an additional four or six cycles of adjuvant CAPOX chemotherapy.
  Interventions: Drug: Tislelizumab; Drug: Oxaliplatin; Drug: Capecitabine
- CAPOX chemotherapy (Placebo Comparator): Patients in the experimental group underwent two or four cycles of preoperative CAPOX combined with placebo. Patients assessed as suitable for R0 resection by imaging underwent radical colectomy. Following surgery, all patients in both groups completed an additional four or six cycles of adjuvant CAPOX chemotherapy.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Tislelizumab — 200 mg on Day 1 every 3 weeks and repeat for 2 or 4 cycles. The incidence of adverse events with Tislelizumab is relatively low. The Tislelizumab dose adjustment was implemented according to the prescribing information.
  Other Names: Baizean
  Arms: CAPOX combined with Tislelizumab
Drug: Oxaliplatin — Oxaliplatin 130mg/m2 on Day 1 every 3 weeks and repeat for 2 or 4 cycles. The dose reduction protocol for oxaliplatin-induced toxicity was implemented according to the study in British Journal of Cancer (2018) 118:1322-1328.
  Other Names: Eloxatin
Drug: Capecitabine — Oral Capecitabine 1000 mg/m2 twice daily combined with oxaliplatin chemotherapy from Day 1 to Day 14 every 3 weeks and repeat for 2 or 4 cycles. The dose reduction protocol for capecitabine-induced toxicity was implemented according to the study in British Journal of Cancer (2018) 118:1322-1328.
  Other Names: Xeloda

SUMMARY:
Building on earlier exploratory work, this study further designs a multi-institutional, prospective, randomized clinical trial to evaluate the efficacy and safety of the combination therapy of the immune checkpoint inhibitor Tislelizumab with CAPOX for neoadjuvant treatment in high-risk locally advanced MSS-type colorectal cancer, as well as its impact on patient outcomes. This study aims to provide new evidence for the clinical practice of treating MSS-type colorectal cancer.

DETAILED DESCRIPTION:
Patients were randomly assigned to either the experimental group, receiving neoadjuvant therapy with Tislelizumab combined with CAPOX, or the control group, receiving neoadjuvant CAPOX chemotherapy alone. Patients in the experimental group underwent four cycles of neoadjuvant CAPOX chemotherapy plus Tislelizumab prior to surgery. Patients in the control group received four cycles of neoadjuvant CAPOX chemotherapy alone. Patients deemed eligible for R0 resection based on radiographic assessment proceeded to radical colorectal cancer surgery. Following surgery, patients in both groups were to complete an additional four cycles of CAPOX chemotherapy. We compared and analyzed the short- and long-term clinical outcomes between the Tislelizumab plus CAPOX regimen and CAPOX alone for the treatment of microsatellite stable (MSS)-type high-risk locally advanced colon cancer (stages T4NanyM0 or TanyN+M0).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and ≤75 years old.
* Pathologically diagnosed MSS ((confirmed by microsatellite stable detection or next-generation target sequencing) or (confirmed by immunohistochemistry)) colon adenocarcinoma.
* The lower edge of the tumor is more than 12cm from the anus as measured by colonoscopy and the lower edge of the tumor cannot be directly palpated during rectal examination.
* Enhanced CT stage T4 or T1-4 N+ without multiple primary tumors or distant metastasis.
* The Eastern Cooperative Oncology Group physical status score is 0-1.
* Life expectancy is expected to be more than 1 year.
* First diagnosis, no previous anti-tumor treatment received, and no chemotherapy contraindications.
* Appropriate organ function is defined as follows: Hemoglobin level ≥ 60g/L, Neutrophil count ≥ 1.5×10^9/L, Platelet count ≥ 75×10^9/L, Serum total bilirubin ≤ 1.5× the upper limit of normal (UNL), Aspartate aminotransferase (AST) ≤ 2× UNL, Alanine aminotransferase (ALT) ≤ 3× UNL, Serum creatinine ≤ 1.5× UNL.
* Informed consent, able to understand the study protocol and willing to participate in the study, and will provide written informed consent.

Exclusion Criteria:

* Enhanced CT stage (T1-3N0M0)
* Multifocal colorectal cancer.
* CT or MRI in the mid-sagittal plane shows that the lower border of the tumor is below the line connecting the sacrococcygeal promontory and the upper border of the pubic symphysis.
* Tumor obstruction or high risk of obstruction, bleeding, and/or perforation requiring emergency surgery or stent placement.
* Cannot tolerate chemotherapy or immunotherapy, such as but not limited to bone marrow suppression.
* History of malignant tumors, except for basal cell carcinoma, papillary thyroid carcinoma, and various in situ cancers.
* Acute exacerbation of important organ diseases (such as but not limited to chronic obstructive pulmonary disease, coronary heart disease, and renal insufficiency) and/or severe acute infectious diseases (such as but not limited to hepatitis, pneumonia, and myocarditis), American Society of Anesthesiologists score > 3 points.
* Mental disorders, illiteracy, or language communication barriers that prevent the understanding of the study protocol.
* Peripheral sensory neuropathy, unable to receive oxaliplatin-based chemotherapy.
* Continuous use of glucocorticoids for more than 3 days within 1 month prior to signing the informed consent form, or having comorbidities requiring the use of glucocorticoid therapy.
* Unable to undergo enhanced CT examination
* Pregnancy or lactation.
* Refused to participate in this study.
* Other situations in which the researcher deems unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | 3-5 days of postoperative pathological examination
  the proportion of tumor regression grades 0 (TRG0, disappearance of tumor cells) in the pathological specimens of surgically resected tumors.

SECONDARY OUTCOMES:
R0 resection | 3-5 days of postoperative pathological examination
  the rate of a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed.
Disease-free survival (DFS) | From date of the patient signs the informed consent form until the date of earliest occurrence of the patient's tumor recurrence or death, whichever came first, assessed up to 36 months.
  3-year disease-free survival
Overall survival (OS) | From the date of the patient signs the informed consent form until the date of the patient's death, assessed up to 36 months.
  3-year overall survival
Adverse events (AEs) | up to half a year
  the rate of adverse events
Immune-related adverse events (irAEs) | up to half a year
  the rate of immune-related adverse events
Surgical complication | From the day of surgery to 30 days after the operation, including intraoperative and postoperative complications.
  the rate of surgical complication during or after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Sen Zhang, Study Director — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China